CLINICAL TRIAL: NCT00171574
Title: Antiproteinuric Effect of Valsartan, Lisinopril and Valsartan Plus Lisinopril in Non-diabetic and Diabetic Renal Disease: a Randomized, Double Blind, Parallel Group, Controlled Trial With 5 Months Follow-up
Brief Title: Antiproteinuric Effect of Valsartan and Lisinopril
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAL489AES13
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Hypertension; Diabetic Nephropathy
Keywords: valsartan; lisinopril; antiproteinuric; diabetic nephropathy
MeSH Terms: conditions — Hypertension; Diabetic Nephropathies | interventions — Valsartan; Hydrochlorothiazide; Lisinopril

INTERVENTIONS:
Drug: Valsartan
Drug: Valsartan plus HCTZ
Drug: Lisinopril

SUMMARY:
Title: Antiproteinuric effect of valsartan, lisinopril and valsartan versus lisinopril in non-diabetic and diabetic renal disease: a randomized (3:3:1), double blind, parallel group, controlled trial, 5 months follow-up.

Objective: To evaluate the antiproteinuric effect of high doses of valsartan vs combo treatment in no-diabetic and diabetic patients.

Hypothesis: Combo treatment reduces microalbuminuria, proteinuria and the albumin/creatinin ratio more than monotherapies.

Design: Multicentric, randomized, double blind, parallel group, active controlled.

Dose / regimen Valsartan 320 vs Lisinopril 40 vs Valsartan/lisinopril 160/20

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients aged 18-70 years,
2. Chronic nephropathy, as defined by a serum creatinine concentration of > 3 mg/dL or calculated glomerular filtration rate of > 30 mL/min/1.73 m2.
3. Persistent proteinuria, as defined by urinary protein excretion exceeding 1g/24 h. (for a minimum of three months ).
4. Normotensive and hypertensive patients not adequately controlled with or without treatment (controlled: <125/75 mmHg).
5. Written informed consent to participate in the study prior to any study procedures.

Exclusion Criteria

* Immediate need for renal replacement therapy.
* Treatment resistant oedema.
* Need for treatment with corticosteroids, non-steroidal anti-inflammatory drugs, or immunosuppressive drugs.
* Proteinuria greater than 10g /24h and/or hypoalbuminaemia less than 28g/L.
* Renovascular hypertension
* Malignant hypertension
* MI, cerebrovascular accident within last year, severe peripheral vascular disease, CHF, chronic hepatic disease.
* Angiotensin converting enzyme inhibitors and angiotensin II receptors blockers within one month prior to randomization.
* A serum creatinine concentration >265 ümol/L

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2004-11; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in urine protein excretion after 20 weeks

SECONDARY OUTCOMES:
Change from baseline in a laboratory measure of kidney function after 20 weeks
Change from baseline in systolic blood pressure after 20 weeks
Change from baseline in diastolic blood pressure after 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Basel, Switzerland